CLINICAL TRIAL: NCT02588001
Title: Japanese Research for Patients With Non-metastatic Castration Resistant Prostate Cancer - Enzalutamide
Acronym: JCASTRE-Zero
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Kagawa University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIGU1506; UMIN000018964 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enzalutamide Group (Experimental)
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — All patients will receive enzalutamide 160 mg (four 40 mg capsules) orally once daily. The treatment will be started at Visit 0 within one week after enrollment. Visit 1 is at 2 weeks after the treatment started; clinical assessments are conducted on adverse events and the Japanese version of the Functional Assessment of Cancer Therapy-Prostate (FACT-P) scales. Patients who are considered to be adequate by the investigator can continue the treatment with 12-week cycle visit (counted from initial dose) until patients meet withdrawal criteria. Patients will be followed up at 2 and 3 years after enrollment and at 3 years after the last participant enrollment.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of enzalutamide in patients with non-metastatic castration resistant prostate cancer. The total duration of the study will be 5 years. All patients will receive enzalutamide 160 mg (four 40 mg capsules) orally once daily. The treatment will be started at Visit 0 within one week after enrollment. Visit 1 is at 2 weeks after the treatment started; clinical assessments are conducted on adverse events and the Japanese version of the Functional Assessment of Cancer Therapy-Prostate (FACT-P) scales. Patients who are considered to be adequate by the investigator can continue the treatment with 12-week cycle visit (counted from initial dose) until patients meet withdrawal criteria. Patients will be followed up at 2 and 3 years after enrollment and at 3 years after the last participant enrollment. The end of the study is defined as follow-up assessment date at 3 years after the last participant enrollment. Patients will primarily be assessed by prostate-specific antigen (PSA) progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed prostate cancer
2. Patients with history of radical prostatectomy or radiation therapy for radical treatment
3. Patients who receive continuous androgen deprivation therapy using both gonadotropin-releasing hormone (GnRH) agonist and antagonist, or using surgical castration
4. Patients with serum testosterone 1.73 nmol/L (0.50 ng/dL) or less
5. Patients with history of bicalutamide or flutamide at any time after first recurrence confirmed since radical treatment completed
6. Patients with 3 increased PSA test results which measured consecutively at least one week apart during androgen deprivation therapy
7. Patients with serum PSA 1 micrograms/L (1 ng/mL) or more
8. Patients with no confirmed remote metastasis after diagnosis of prostate cancer (excluding lymph nodes metastasis with a minor axis of less than 15 mm which considered to be nonmeasurable in the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1)
9. Patients with asymptomatic prostate cancer
10. Patients with the Eastern Cooperative Oncology Group (ECOG) performance status 0-1
11. Patients with life expectancy of at least 12 months
12. Patients who have signed written informed consent to participate in this study

Exclusion Criteria:

1. Patients with history of any chemotherapy (including estramustine phosphate sodium hydrate (JAN)) or treatment with enzalutamide or abiraterone acetate
2. Patients with history of steroid usage as treatment for prostate cancer
3. Patients with history of 5-alpha-reductase inhibitor, estrogen or steroidal antiandrogen within past 4 weeks prior to initial administration of enzalutamide
4. Patients with history of malignant tumor other than prostate cancer within past 3 years
5. Patients with history of seizure or predisposing disease of seizure
6. Patients with severe liver dysfunction
7. Patients with a previous history of hypersensitivity to any component of drugs which will be administered in this study
8. Patients who considered to be inappropriate for the study participation by the investigator.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
PSA-progression-free survival (PSA-PFS) | 6 years
  Prostate specific antigen (PSA) progression-free survival is defined as time from date of initial dose until the date of first confirmed PSA progression (an increase in PSA of >= 25% and >= 2 ng/ml above the nadir after initial dose) or date of death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival (OS) | 6 years
  OS is defined as time from date of initial dose until date of death from any cause.
Progression-free survival (PFS) | 6 years
  PFS is defined as time from date of initial dose until the date of first confirmed progression or date of death from any cause, whichever comes first.
Metastasis free survival (MFS) | 6 years
  MFS is defined as time from date of initial dose until the date of first metastasis which confirmed by computed tomography (CT) and bone scintigraphy.
Time-to-PSA-progression (TTPP) | 6 years
  TTPP is defined as time from date of initial dose until the date of first confirmed PSA progression (an increase in PSA of >= 25% and >= 2 ng/ml above the nadir after initial dose).
PSA response rate | At week 2, and every 12 weeks for up to 6 years after initial dose
  PSA response rate is defined as ratio of patients who have an decrease in PSA of >= 50% above baseline, compared to PSA levels at week 2, every 12 weeks for up to 5 years after initial dose.
Time to first use of chemotherapy (TFC) | 6 years
  TFC is defined as time from date of initial dose until the date of first additional chemotherapy started for prostate cancer.
QOL assessment using Japanese version of the FACT-P scales | Baseline, week 2, week 60, at withdrawal of treatment and at end of treatment for up to 6 years
  Quality of life (QOL) is assessed on both total scores and each domain scores using Japanese version of the Functional Assessment of Cancer Therapy-Prostate (FACT-P) scales at baseline, week 2, week 60, withdrawal of treatment and at the end of treatment for up to 5 years.
Medication adherence (dosage) | 6 years
  Medication adherence is assessed in dosage of enzalutamide.
Medication adherence (duration) | 6 years
  Medication adherence is assessed in duration of enzalutamide.
Medication adherence (ratio) | 6 years
  Medication adherence is assessed in dosage rate of enzalutamide which is classfied into 3 categories: 1) >=80%, 2) >= 50% to < 80%, and 3) < 50%.
Safety assessment on the incidence and severity of adverse events using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Mikio Sugimoto, MD, Ph.D., Principal Investigator — Kagawa University
Locations (4):
- Japan (4):
  - Kagawa University Faculty of Medicine, Kita-gun, Kagawa-ken
  - University of Miyazaki Faculty of Medicine, Miyazaki, Miyazaki
  - Tokyo Medical Center, Meguro-ku, Tokyo
  - The Jikei university school of medicin, Minato-ku, Tokyo